CLINICAL TRIAL: NCT05459532
Title: This is a Multi-centre, Double-blind, Phase 3 Study to Observe the Effectiveness, Safety, and Tolerability of Molnupiravir 800 mg Administered 12-hourly for Five Days to Adult Patients With Mild COVID-19 at the Time of Enrolment Who Are at Risk of Progression to Severe Disease, Compared to a Placebo. Patients With Recent Onset of COVID-19 Symptoms Will be Screened to Assess Eligibility for Enrolment. Confirmation of SARS-CoV-2 Infection Will be Performed Through Rapid Antigen Detection Using the LumiraDx Point of Care Diagnostic Platform.
Brief Title: A Randomised, Multi-centre, Double-blind, Phase 3 Study to Observe the Effectiveness, Safety and Tolerability of Molnupiravir Compared to Placebo Administered Orally to High-risk Adult Outpatients With Mild COVID-19 Receiving Local Standard of Care in South Africa
Acronym: CoTeT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Witwatersrand, South Africa (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Professor Francois Venter, Head: Clinical Research, University of Witwatersrand, South Africa
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EZ-SS-029
Record Dates: First submitted 2022-07-13; First posted 2022-07-15 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — molnupiravir

STUDY DESIGN:
Intervention Model Description: Molnupiravir is a broad-spectrum antiviral that is an orally bioavailable prodrug of the nucleoside analogue NHC. NHC distributes into cells where it is phosphorylated to form the pharmacologically active NHC-TP. NHC-TP acts by a mechanism known as viral error catastrophe. NHC-TP incorporation into viral RNA by the viral RNA polymerase, results in an accumulation of errors in the viral genome leading to inhibition of replication.
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monulpiravir (Experimental): Eligible participants will be randomised in a 1:1 manner to receive either molnupiravir 800 mg orally approximately 12-hourly for five days or a placebo for the equivalent amount of time.
  Interventions: Drug: Molnupiravir 200 mg
- Placebo (Placebo Comparator): Eligible participants will be randomised in a 1:1 manner to receive either molnupiravir 800 mg orally approximately 12-hourly for five days or a placebo for the equivalent amount of time.
  Interventions: Drug: Molnupiravir 200 mg

INTERVENTIONS:
Drug: Molnupiravir 200 mg — The drug is orally bioavailable (and is indicated for treatment of mild to moderate COVID-19 in adults with a positive SARS-COV-2 diagnostic test and who have at least one risk factor for developing severe illness. The recommended dose is 800 mg (four 200 mg capsules) taken orally 12-hourly for five days, and should be administered as soon as possible after diagnosis of COVID-19 has been made and within five days of symptom onset.

SUMMARY:
This is a multi-centre, double-blind, phase 3 study to observe the effectiveness, safety, and tolerability of molnupiravir 800 mg administered 12-hourly for five days in adult patients with mild COVID-19 at the time of enrolment, who are at risk of progression to severe disease, compared to a placebo.

DETAILED DESCRIPTION:
This is a multi-centre, double-blind, phase 3 study to observe the effectiveness, safety, and tolerability of molnupiravir 800 mg administered 12-hourly for five days in adult patients with mild COVID-19 at the time of enrolment, who are at risk of progression to severe disease, compared to a placebo.

Patients with recent onset of COVID-19 symptoms will be screened to assess eligibility for enrolment. Confirmation of SARS-CoV-2 infection will be performed through rapid antigen detection using the LumiraDx point of care diagnostic platform. Approximately 4000 eligible patients will be enrolled and will be randomised in a 1:1 manner to start treatment with either molnupiravir or a placebo on the same day. Patients will record their symptoms (through a self-administered questionnaire) and self-observed vital signs daily for 10 days from the time of enrolment and will be contacted by study team personnel on Days 3, 6 and 10 to monitor their well-being. Adverse event and concomitant medication data will be collected. A final end-of-study follow-up visit will be conducted on Day 29.

An independent Data and Safety Monitoring Board (DSMB) will be convened for this study with expertise in COVID-19 or respiratory viruses, and emerging epidemics. The purpose of the DSMB is to monitor the study for safety and operational futility.

In addition to the usual, regular, required reporting to SAHPRA, the investigator anticipates that additional reporting will be required by the Clinical Trials Committee, noting the severity of the 3rd and 4th waves, the level of ''breakthrough'' infections in the context of high background comorbidities, and the urgent interest in this class of drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written or electronic informed consent prior to any study-specific procedure.
2. Age ≥50 at the time of signing the informed consent form.
3. Women of reproductive potential must have a negative pregnancy test at screening and be using a highly effective method of contraception. Highly effective methods of contraception
4. A male participant must wear a condom when engaging in any activity that allows for passage of ejaculate to another while taking the investigational product. Male participants should also be advised of the benefit for a female partner to use a highly effective method of contraception as condom may break or leak.
5. Self-reported symptoms of COVID-19 with onset no more than five days prior to screening informed consent including at least one of, fever or chills, cough, sore throat, rhinorrhoea or rhinitis or sinusitis, shortness of breath, headache, myalgia, new onset anosmia or ageusia, nausea, diarrhoea, or extreme fatigue, or other symptoms recognized in local and international guidelines as typical of mild COVID-19.
6. SARS-CoV-2 infection confirmed through a positive LumiraDx rapid antigen test on the day of screening or a positive RT-PCR within two days prior to screening.
7. Participant is at high risk for progression to severe COVID-19, this defined as either:

   1. Age ≥50 with at least one of the following background or medical conditions: diabetes mellitus, obesity (BMI 30 kg/m2), hypertension, HIV, active or previous TB.
   2. Age ≥65
8. Participant agrees to comply with study procedures, including the completion of a daily diary for 10 days from the time of enrolment, and to be available for study contacts and visits.

   -

Exclusion Criteria:

1. Pregnant or breastfeeding women, or women planning/desiring to become pregnant during the 28 days following enrolment into the study.
2. Duration of self-reported symptoms of COVID-19 for more than five days prior to screening.
3. Signs of respiratory distress or severe disease prior to enrolment, including:
4. Inability/unlikely to be in the study area for the duration of the 28-day follow-up period.
5. Inability to tolerate oral medications.
6. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the safety of the patient or the objectives of the study. The Investigator should make this determination in consideration of the volunteer's medical history.
7. The volunteer is assessed to be clinically unstable in the Investigator's opinion.
8. Participation in another investigational study involving an investigational product within 30 days, or 5 half-lives, whichever is longer, prior to screening.
9. Personnel (e.g., investigator, sub-investigator, research assistant, pharmacist, study coordinator or anyone mentioned in the delegation log) directly involved in the conduct of the study.
10. Any physical, mental, or social condition, drug/alcohol use, history of illness or laboratory abnormality that, in the Investigator's judgment, might jeopardise the safety of the patient in the context of this study, or might interfere with study procedures or the ability of the subject to adhere to and complete the study. The Investigator should make this determination in consideration of the volunteer's medical history.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the effectiveness of molnupiravir compared to placebo in preventing severe disease progression in adults with mild COVID-19 | 29 Days
  Combination of incidence of COVID-19-related hospitalisation (24 hours of care in a hospital or similar acute care facility) and COVID-19-related mortality to Day 29
To evaluate the safety of molnupiravir in adults with mild COVID-19 | 29 Days
  Adverse events (including serious adverse events and adverse drug reactions)
To evaluate the safety of molnupiravir in adults with mild COVID-19 | 29 Days
  Self-assessed vital signs to Day 10

SECONDARY OUTCOMES:
To facilitate same-day COVID-19 diagnosis and treatment initiation in adults with mild COVID-19 and comorbid conditions | 29 Days
  Proportion of enrolled patients for whom diagnosis and same day treatment initiation was facilitated through use of a LumiraDx™ rapid antigen test
To assess the tolerability of molnupiravir in adults with mild COVID-19 | 29 Days
  Severity of adverse events
To assess the tolerability of molnupiravir in adults with mild COVID-19 | 29 Days
  Adverse event-related study drug discontinuations
To describe time to symptom resolution in adults with mild COVID-19 treated with molnupiravir compared to placebo | 29 Days
  Time to sustained resolution of symptoms as reported in the Flu-PRO© Plus
To evaluate maximum COVID-19 disease severity in adults treated with molnupiravir compared to placebo | 29 Days
  Maximum score on the WHO Clinical Progression Scale from Day 1 to Day 29
To evaluate the relationship between effectiveness of molnupiravir and time between onset of symptoms and initiation of treatment | 29 Days
  Number of days from symptom onset to initiation of treatment
To evaluate the relationship between effectiveness of molnupiravir and time between onset of symptoms and initiation of treatment | 29 Days
  Incidence of hospitalisation (24 hours of care in a hospital or similar acute care facility) and/or death to Day 29 in patients with co-morbid conditions
To evaluate the relationship between effectiveness of molnupiravir and time between onset of symptoms and initiation of treatment | Day 1 to Day 10 and Day 29
  Time to sustained resolution of symptoms as reported in the Flu-PRO Plus
To evaluate the relationship between effectiveness of molnupiravir and time between onset of symptoms and initiation of treatment | Day 0, 3, 6, 10, 29
  Maximum score on the WHO Clinical Progression Scale from Day 1 to Day 29. On a scale of 0 to 10 (0 being uninfected and 10 being worse/death)
To describe adherence to a 5-day course of molnupiravir in adults with mild COVID-19 | 29 Days
  Proportion of patients completing the course of molnupiravir as prescribed
To describe the utilisation of health care services by adults with mild COVID-19 treated with molnupiravir compared to placebo | 29 Days
  Rate of hospital, emergency facility, clinic, health care practitioner or home visits to Day 29
To report the incidence and outcome of pregnancies in female participants who received molnupiravir | 29 Days
  Incidence of pregnancy in female participants to Day 29
To report the incidence and outcome of pregnancies in female participants who received molnupiravir | Once
  20-week gestational age ultrasound findings
To report the incidence and outcome of pregnancies in female participants who received molnupiravir | Throughout the pregnancy
  Pregnancy complications
To report the incidence and outcome of pregnancies in female participants who received molnupiravir | Once
  Pregnancy outcome
To report the incidence and outcome of pregnancies in female participants who received molnupiravir | Once
  Infant wellbeing to three months of age

CONTACTS AND LOCATIONS:
Overall Officials: Francois WD Venter, Study Director — Ezintsha, Faculty of Health Sciences University of the Witwatersrand
Locations (4):
- South Africa (4):
  - Nelson Mandela Academic Clinical Research Unit (NeMACRU), Umtata, Eastern Cape
  - Sunnyside Office Park, Johannesburg, Gauteng
  - Nelson R. Mandela School of Medicine 3rd Floor, K-RITH Tower Building, Durban, KwaZulu-Natal
  - The Aurum Institute: Gavin J Churchyard Legacy Centre Klerksdorp Clinical Research Centre, Klerksdorp, North West

IPD SHARING:
Plan to Share IPD: Yes
The data that will be shared is all of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: Immediately following publication
Access Criteria: Anyone who wishes to access the data

DOCUMENTS (2):
  • Study Protocol (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/32/NCT05459532/Prot_000.pdf
  • Informed Consent Form (2022-05-30): https://cdn.clinicaltrials.gov/large-docs/32/NCT05459532/ICF_001.pdf